CLINICAL TRIAL: NCT00162578
Title: Vancomycin Concentration in Cerebrospinal Fluid During Pneumococcal Meningitis Treated With Dexamethasone
Brief Title: Vancomycin Concentration in Cerebrospinal Fluid During Pneumococcal Meningitis
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Other Study IDs: LMR4
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-07

CONDITIONS: Pneumococcal Meningitis
Keywords: pneumococcal meningitis; intensive care unit; vancomycin; dexamethasone; drug diffusion in cerebrospinal fluid
MeSH Terms: conditions — Meningitis, Pneumococcal

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Adding vancomycin to the antibiotic regimen is recommended for the treatment of pneumococcal meningitis in adults. Use of dexamethasone as adjunct therapy has proved to reduce mortality and neurologic sequelae in adult patients with pneumococcal meningitis. However, use of dexamethasone may impair penetration of vancomycin in cerebrospinal fluid. In a purely observational manner, we thought to measure blood and CSF concentrations of vancomycin in adult patients with pneumococcal meningitis, treated with vancomycin, third-generation cephalosporin and dexamethasone.

DETAILED DESCRIPTION:
Because of a considerable increase in streptococcus pneumoniae meningitis with penicillin nonsusceptible strains, it is now largely recommended to add vancomycin to the third-generation cephalosporin antibiotic regimen. It has also been recently shown that use of dexamethasone reduces mortality and unfavorable outcome in adults with pneumococcal meningitis. However, concern has arisen, that dexamethasone may impair penetration of vancomycin in cerebrospinal fluid.

We therefore thought to measure in a purely observational study, blood and CSF vancomycin concentrations in adult patients with pneumococcal meningitis hospitalized in medical intensive care unit that received third-generation cephalosporin, vancomycin and dexamethasone. The aim of the study was to observe whether or not sufficient concentrations of vancomycin could be measured in the CSF despite the concomitant use of dexamethasone. Patients were cared for in a perfectly routine manner. There was no randomization. All patients received routine, recommended care (IDSA guidelines). There was no invasive procedure. Dexamethasone was administered according to the de Gans study (NEJM 2002). In these patients with severe meningitis, a second lumbar puncture was performed as recommended(IDSA Guidelines, CID 2004). At the same time, peripheral blood was taken. In both samples, vancomycin concentration was determined.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 yr) with suspicion of pneumococcal meningitis requiring intensive care unit

Exclusion Criteria:

* Allergy to one of the antibiotics used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2002-12; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Didier DREYFUSS, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Service de Réanimation Médicale, CHU Louis Mourier, Colombes
  - Service de Réanimation Médicale, CHU Bichat, Paris
  - Service de Réanimation Médicale, CHI Poissy-St-Germain, Poissy

REFERENCES:
- [Background] Tunkel AR, Hartman BJ, Kaplan SL, Kaufman BA, Roos KL, Scheld WM, Whitley RJ. Practice guidelines for the management of bacterial meningitis. Clin Infect Dis. 2004 Nov 1;39(9):1267-84. doi: 10.1086/425368. Epub 2004 Oct 6. No abstract available. PMID 15494903
- [Background] de Gans J, van de Beek D; European Dexamethasone in Adulthood Bacterial Meningitis Study Investigators. Dexamethasone in adults with bacterial meningitis. N Engl J Med. 2002 Nov 14;347(20):1549-56. doi: 10.1056/NEJMoa021334. PMID 12432041
- [Background] Auburtin M, Porcher R, Bruneel F, Scanvic A, Trouillet JL, Bedos JP, Regnier B, Wolff M. Pneumococcal meningitis in the intensive care unit: prognostic factors of clinical outcome in a series of 80 cases. Am J Respir Crit Care Med. 2002 Mar 1;165(5):713-7. doi: 10.1164/ajrccm.165.5.2105110. PMID 11874820
- [Background] Viladrich PF, Gudiol F, Linares J, Pallares R, Sabate I, Rufi G, Ariza J. Evaluation of vancomycin for therapy of adult pneumococcal meningitis. Antimicrob Agents Chemother. 1991 Dec;35(12):2467-72. doi: 10.1128/AAC.35.12.2467. PMID 1810180
- [Derived] Ricard JD, Wolff M, Lacherade JC, Mourvillier B, Hidri N, Barnaud G, Chevrel G, Bouadma L, Dreyfuss D. Levels of vancomycin in cerebrospinal fluid of adult patients receiving adjunctive corticosteroids to treat pneumococcal meningitis: a prospective multicenter observational study. Clin Infect Dis. 2007 Jan 15;44(2):250-5. doi: 10.1086/510390. Epub 2006 Dec 15. PMID 17173226